CLINICAL TRIAL: NCT00703651
Title: Immunogenicity of Two Dosages of Inactivated, Split-Virion Influenza Vaccine Administered by Intradermal Route in Comparison With Intramuscular Vaccination With Vaxigrip® in Adults
Brief Title: Study of Inactivated, Split-Virion Influenza Vaccine Administered by Intradermal Route Versus Vaxigrip® in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GID02
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Influenza; Orthomyxoviridae Infection; Myxovirus Infection
Keywords: Influenza; Orthomyxoviridae Infection; Inactivated, Split-virion influenza vaccine; Intradermal injection; Adults.
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections | interventions — vaxigrip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Biological: Inactivated, split-virion influenza vaccine
- 2 (Experimental)
  Interventions: Biological: Inactivated, split-virion influenza vaccine
- 3 (Active Comparator)
  Interventions: Biological: Inactivated, split-virion influenza vaccine

INTERVENTIONS:
Biological: Inactivated, split-virion influenza vaccine — 0.1 mL, ID. 1 injection/year for 3 years
  Arms: 1
Biological: Inactivated, split-virion influenza vaccine — 0.1 mL, ID. 1 injection/year for 3 years.
  Arms: 2
Biological: Inactivated, split-virion influenza vaccine — 0.5 mL, IM. 1 injection/year for 3 years
  Other Names: Vaxigrip®
  Arms: 3

SUMMARY:
This is a follow-up of a previous dose-ranging study aimed at investigating 2 doses of the trivalent inactivated split virion influenza vaccine when administered by intradermal route with that of the current pharmaceutical presentation administered by intramuscular route.

Primary Objective:

To assess the immunogenicity of two pharmaceutical presentations of the trivalent inactivated split virion influenza vaccine 21 days after a single injection in subjects aged 18 to 57 years.

Secondary Objective:

To evaluate the safety profile during the 21-day period following each vaccination in each study group

DETAILED DESCRIPTION:
This is an open (for the administration route) and double-blind (only for the two dosages administered at year 0 by using the investigational administration route) randomized trial conducted in subjects aged 18 to 60 years. The subjects will receive three vaccine injections at 1-year interval.

ELIGIBILITY:
Inclusion Criteria :

* Subject aged between 18 and 57 years (i.e., less than 60 at the last vaccination)
* For woman of child-bearing potential, negative urine pregnancy test at V#01
* Use of effective contraception prior to and during the trial
* Subject available during the trial period
* Subject able to read and understand the informed consent form
* Informed consent form signed and dated by the subject prior to any protocol-required intervention (and Visit 05 and Visit 07, respectively).

Exclusion Criteria :

* Self-reported allergy to egg proteins, chick proteins, or any of the constituents of the vaccine, in particular, neomycin, formaldehyde, and octoxinol 9
* Acute febrile disease within the 72 hours preceding V#01, or axillary temperature >37.5°C the day of inclusion, prior to vaccination (>37.0°C Czech Republic)
* Subject with an aggravation of existing chronic illness (heart disease, respiratory disease, etc.)
* Vaccination against influenza within the 6 months preceding V#01
* Any vaccination within the 28 days preceding V#01 or scheduled between V#01 and V#02
* Breast-feeding
* Immunosuppressive therapy including long term systemic corticotherapy (20 mg/day of prednisolone or equivalent for >2 weeks) or cancer therapy within the month preceding V#01 or ongoing
* Immunoglobulin injection within the 3 months preceding V#01
* Subject taking part or planned to take part in another clinical trial (3 months before and through the trial duration)
* Subject having received extracted pituitary hormones
* Subjects who participated in the GID01 study (Lithuanian centers)

Ages: 18 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1150 (Actual)
Dates: Start 2003-09; Primary Completion 2006-05 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of Inactivated, Split-Virion Influenza Vaccine. | 21days post-vaccination
To provide information concerning the safety of Inactivated, Split-Virion Influenza Vaccine | 21 days post-vaccination and entire study duration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasterur Inc
Locations (8):
- Belgium (5):
  - Gribomont
  - Kraainem
  - Linkebeek
  - Molenbeek
  - Thuin
- Hradec Králové, Czechia
- Lithuania (2):
  - Kaunas
  - Vilnius

REFERENCES:
- [Derived] Beran J, Ambrozaitis A, Laiskonis A, Mickuviene N, Bacart P, Calozet Y, Demanet E, Heijmans S, Van Belle P, Weber F, Salamand C. Intradermal influenza vaccination of healthy adults using a new microinjection system: a 3-year randomised controlled safety and immunogenicity trial. BMC Med. 2009 Apr 2;7:13. doi: 10.1186/1741-7015-7-13. PMID 19341446
- See also: Related Info — http://www.sanofipasteur.com